CLINICAL TRIAL: NCT02667444
Title: A Phase 3 Multi-Center, Randomized, Double-Blinded, Vehicle-Controlled, Parallel Group Study Comparing the Efficacy, Tolerability and Safety of Once Daily SB204 and Vehicle Gel in the Treatment of Acne Vulgaris
Brief Title: P3 Study Comparing Once Daily SB204 and Vehicle Gel in Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC302
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB204 4% (Experimental): SB204 4% topically once daily
  Interventions: Drug: SB204 4%
- Vehicle Gel (Placebo Comparator): Vehicle Gel topically once daily
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: SB204 4% — Applied topically once daily
  Other Names: NVN1000
  Arms: SB204 4%
Drug: Vehicle Gel — Applied topically one daily
  Other Names: Placebo
  Arms: Vehicle Gel

SUMMARY:
This is a 12 week, multi-center, double-blinded, randomized, vehicle-controlled, parallel group, study to be conducted in approximately 1300 subjects with acne vulgaris in the US.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled study in subjects with moderate to severe acne. Subjects who satisfy the entry criteria will be randomized to SB204 4% QD or Vehicle Gel QD in a 1:1 ratio. Efficacy assessments will include Investigator Global Assessments (IGA) and inflammatory and non-inflammatory lesion counts. Subjects will return for post-Baseline evaluation at Weeks 2, 4, 8, and 12/Early Termination (ET).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe acne
* Minimum of 25 and no more than 70 non-inflammatory lesions (open and closed comedones) on the face
* Minimum of 20 and no more than 40 inflammatory lesions (papules and pustules)

Exclusion Criteria:

* Women of child-bearing potential who are pregnant, nursing, considering becoming pregnant
* Any dermatologic condition that could interfere with clinical evaluations including severe, recalcitrant cystic acne

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1330 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Study Chair — Novan, Inc.
Locations (55):
- United States (55):
  - CIL #214, Birmingham, Alabama
  - CIL #218, Mobile, Alabama
  - CIL #189, Phoenix, Arizona
  - CIL #139, Cerritos, California
  - CIL #216, Chula Vista, California
  - CIL #181, Encino, California
  - CIL #174, Huntington Beach, California
  - CIL #213, La Mesa, California
  - CIL #190, Sacramento, California
  - CIL #111, San Diego, California
  - CIL #195, Santa Ana, California
  - CIL #119, Santa Monica, California
  - CIL #158, Bradenton, Florida
  - CIL #208, Hialeah, Florida
  - CIL #142, Miami, Florida
  - CIL #170, Miami Lakes, Florida
  - CIL #204, Miami Springs, Florida
  - CIL #185, Ormond Beach, Florida
  - CIL #110, Pinellas Park, Florida
  - CIL #227, Sanford, Florida
  - CIL #176, St. Petersburg, Florida
  - CIL #152, Tampa, Florida
  - CIL #144, Tampa, Florida
  - CIL #116, Newnan, Georgia
  - CIL #143, Savannah, Georgia
  - CIL #175, New Albany, Indiana
  - CIL #191, Overland Park, Kansas
  - CIL #228, Louisville, Kentucky
  - CIL #194, Richmond, Kentucky
  - CIL #219, Monroe, Louisiana
  - CIL #145, Boston, Massachusetts
  - CIL #155, Bay City, Michigan
  - CIL #220, St Louis, Missouri
  - CIL #148, Norfolk, Nebraska
  - CIL #206, Omaha, Nebraska
  - CIL #202, Morristown, New Jersey
  - CIL #197, New York, New York
  - CIL #196, Charlotte, North Carolina
  - CIL #192, Raleigh, North Carolina
  - CIL #221, Salisbury, North Carolina
  - CIL #169, Cincinnati, Ohio
  - CIL #237, Gresham, Oregon
  - CIL #137, Broomall, Pennsylvania
  - CIL #147, Hershey, Pennsylvania
  - CIL #178, Philadelphia, Pennsylvania
  - CIL #160, Austin, Texas
  - CIL #183, Austin, Texas
  - CIL #184, Bryan, Texas
  - CIL #163, Channelview, Texas
  - CIL #165, Dallas, Texas
  - CIL #167, Houston, Texas
  - CIL #223, Plano, Texas
  - CIL #159, San Antonio, Texas
  - CIL #105, Lynchburg, Virginia
  - CIL #231, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Gel: Vehicle Gel: Applied topically once daily
Period: Overall Study
Arm/Group | SB204 4% | Vehicle Gel
Started | 664 | 666
Completed | 576 | 574
Not Completed | 88 | 92

BASELINE CHARACTERISTICS:
Population: Intent to treat population (ITT): All subjects who were randomized and dispensed study medication, grouped according to the treatment group to which they were assigned at the time of randomization. A total of 1330 subjects were randomized but 3 were withdrawn after randomization and prior to being dispensed study medication (1 subject in the SB204 group and 2 in the Vehicle group).
Groups:
- Total: Total of all reporting groups
Arm/Group | SB204 4% | Vehicle Gel | Total
Number analyzed (Participants) | 663 | 664 | 1327
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (8.52) | 21.8 (8.77) | 21.6 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 411 | 398 | 809
  Male | 252 | 266 | 518
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 202 | 209 | 411
  Not Hispanic or Latino | 461 | 455 | 916
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 43 | 45 | 88
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 158 | 147 | 305
  White | 449 | 457 | 906
  More than one race | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 663 | 664 | 1327
Baseline Investigator Global Assessment [Count of Participants; unit: Participants]
  0--clear | 0 | 0 | 0
  1--almost clear | 0 | 0 | 0
  2--mild | 0 | 0 | 0
  3--moderate | 599 | 587 | 1186
  4--severe | 64 | 77 | 141

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Inflammatory Lesion Counts
Description: The absolute change from Baseline in inflammatory lesion counts was to be assessed on the face only (forehead, right and left cheeks, chin, and nose). Inflammatory lesions included papules, pustules, nodules, and cysts.
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: inflammatory acne lesions
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 663 | 664
inflammatory acne lesions | -13.1 (10.27) | -10.9 (10.81)

2. Primary Outcome: Absolute Change From Baseline in Non-inflammatory Lesion Counts
Description: The absolute change from Baseline in non-inflammatory lesion counts was to be assessed on the face only (forehead, right and left cheeks, chin, and nose). Non-inflammatory lesions included open comedones (blackheads) and closed comedones (whiteheads).
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: non-inflammatory acne lesions
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 663 | 664
non-inflammatory acne lesions | -15.3 (14.30) | -12.7 (16.01)

3. Primary Outcome: Proportion of Subjects With Investigator Global Assessment (IGA) Success at Week 12
Description: Proportion of subjects with Investigator Global Assessment (IGA) Success at Week 12 is defined as an IGA score of 0 or 1 (Clear/Almost Clear) and at least a 2 grade improvement from Baseline. The IGA scale is as follows:
  Grade Description 0 Clear: Clear skin with no inflammatory or non-inflammatory lesions.
  1. Almost clear: Rare non-inflammatory lesions with rare papules (papules may be resolving and hyperpigmented, though not pink-red).
  2. Mild: Some non-inflammatory lesions with no more than a few inflammatory lesions.
  3. Moderate: Up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one nodulocystic lesion.
  4. Severe: Up to many non-inflammatory and inflammatory lesions, but no more than a few nodulocystic lesions
Time Frame: Week 12
Population: Intent to treat (ITT) population; subjects who had Week 12 (study completion) visits.
Measure: Count of Participants; unit: Participants
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 592 | 603
Participants | 120 | 89

4. Secondary Outcome: Percent Change in Inflammatory Lesion Count
Description: The percent change from baseline in inflammatory lesion count
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 663 | 664
Percentage change from baseline | -48.5 (36.36) | -39.2 (38.20)

5. Secondary Outcome: Percent Change in Non-inflammatory Lesion Count
Description: The percent change from baseline in non-inflammatory lesion count
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 663 | 664
Percentage change from baseline | -40.5 (36.35) | -33.1 (39.59)

6. Secondary Outcome: Time to Reduction in Inflammatory Lesion Count
Description: Median time to a 35% reduction (improvement) in inflammatory lesion count (Kaplan-Meier analysis)
Time Frame: Week 12
Population: Intent to treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 485 | 436
Days | 38.0 [31.0 to 56.0] | 56.0 [35.0 to 57.0]

7. Secondary Outcome: Time to Improvement in IGA
Description: Median time to a 2 or more grade improvement in IGA (Kaplan-Meier analysis)
Time Frame: Week 12
Population: Intent to treat (ITT) population--Overall number of participants analyzed = number of participants who achieved a 2 or more grade improvement in their IGA score. This was a Kaplan-Meier analysis; for both the SB204 4% and Vehicle Gel treatment groups, the median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 164 | 124
Days
  25% Quartile | 85.0 [85.0 to 86.0] | 87.0 [86.0 to 91.0]
  50% Quartile (Median) | NA [NA to NA] — The median and 95% CI were not estimable because fewer than 50% of subjects achieved a change of 2 or more in their IGA assessment. | NA [NA to NA] — The median and 95% CI were not estimable because fewer than 50% of subjects achieved a change of 2 or more in their IGA assessment.
  75% Quartile | NA [NA to NA] — The median and 95% CI were not estimable because not enough subjects achieved a change of 2 or more in their IGA assessment. | NA [NA to NA] — The median and 95% CI were not estimable because not enough subjects achieved a change of 2 or more in their IGA assessment.

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the subject signed the informed consent and completed any study assessment until the end of the final study visit, approximately 12 weeks.
Description: Adverse events were collected for all subjects who were randomized and received at least one dose of study medication. Three subjects who were randomized to the Vehicle group received SB204 and per the definition of the Safety Population in the Statistical Analysis Plan, these subjects were analyzed in the SB204 group. Therefore, 666 subjects were in the SB204 group and 661 subjects were in the Vehicle group for analyses of all cause mortality, adverse events and serious adverse events.
Arm/Group | SB204 4% | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/666 | 0/661
Serious Adverse Events (participants affected / at risk) | 1/666 | 3/661
Other Adverse Events (participants affected / at risk) | 49/666 | 25/661
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB204 4% (N=666) | Vehicle Gel (N=661)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorhage (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB204 4% (N=666) | Vehicle Gel (N=661)
Application site pain (General disorders) | 14 | 4
Application site erythema (General disorders) | 10 | 2
Nasopharyngitis (Infections and infestations) | 15 | 18
Headache (Nervous system disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT02667444/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT02667444/SAP_001.pdf